CLINICAL TRIAL: NCT01378806
Title: Children and Parents Partnering Together to Manage Their Weight
Brief Title: Family Partners for Health
Acronym: WEIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Diane Berry, PhD, ANP-BC/Associate Professor, The University of North Carolina at Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-0436; R0100254-05 (Other Grant/Funding Number: NINR); 5-34696 (Other: The University of North Carolina at Chapel)
Record Dates: First submitted 2011-06-02; First posted 2011-06-22 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Overweight; Obesity
Keywords: overweight; obesity; adults; children
MeSH Terms: conditions — Overweight; Obesity | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): A 12-week intensive intervention on nutrition and exercise education and coping skills training (Phase I), 9 months of continued monthly contact (Phase II), and then 6 months on their own.
  Interventions: Behavioral: Nutrition and exercise education and coping skills training

INTERVENTIONS:
Behavioral: Nutrition and exercise education and coping skills training — A 12-week intensive intervention on nutrition and exercise education and coping skills (Phase I), 9 months of continued monthly contact (Phase II), and then 6 months on their own.

SUMMARY:
Young children who are overweight or at risk for overweight are at increased risk for becoming obese as young adults and developing type 2 diabetes and cardiovascular disease. To date, there have been no interdisciplinary interventions that targeted predominantly ethnic minority low-income children and parents and taught them to work together to improve nutrition and exercise. Using a two-group, repeated measures experimental design, this proposed study will test a 12-week intensive intervention on nutrition, exercise and coping skills (Phase I) and 9 months of continued monthly contact (Phase II) to help overweight 2nd, 3rd, and 4th grade children and their parents improve self-efficacy, health behaviors, weight status, and adiposity. The study will take this intervention to the community in which children and parents live, working with four schools in Alamance-Burlington County, NC, and four schools in Wilson County in the early evening. A total of 356 Black, Hispanic, and White children with a BMI >85th percentile and 356 parents with a BMI >25 kg/m2 will be inducted over 3 ½ years and randomized by school to either the experimental or control group. Data will be collected at Time 1 (Baseline), Time 2 (Post Phase I-Intensive Intervention), Time 3 (Post Phase II-Continued Contact), and Time 4 (6-Month Follow-Up). Data collected will include scores on the Health Promoting Lifestyle Profile II in the parents; eating self-efficacy in the children (CATCH) and parents (Eating Self-Efficacy Scale) and exercise self-efficacy in the children (CATCH) and parents (Exercise Self-Efficacy); health behaviors in the children and parents (3 Day 24-Hour Food Recall and 4 Day Accelerometry Measurement); weight status in the children (BMI percentile) and parents (BMI); and adiposity in the children and parents (waist circumference and triceps and subscapular skinfolds). Data analysis will use general linear mixed models to test the hypotheses. Decreasing overweight in children and parents is urgently needed, and helping children and parents to work together to improve their nutrition and exercise patterns by making small lifestyle pattern changes may decrease future health care costs and decrease morbidity and mortality. The knowledge to be gained from this study may provide a foundation for extending this intervention to other Black, Hispanic, and White children and parents in other communities to assist them to manage their weight.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria for children include:

* ability to speak, write, and read in English
* a BMI > 85th percentile for age and gender
* at least one parent or guardian with a BMI >25
* assent and their parent or guardian's consent to their participation

Inclusion criteria for parents or guardians include:

* ability to speak, write, and read in English
* a BMI >25
* a 2nd, 3rd or 4th grade child with a BMI > 85th percentile for age and gender
* reside with the child; and consent to join the study

Exclusion Criteria: Parents and children will be excluded if either has a:

* history of a heart murmur
* congenital heart disease
* family history of sudden death
* history of psychological problems such as claustrophobia that would prevent participation in group classes
* participation in another clinical trial or intervention
* Asians will be excluded since there is a higher level of risk at a lower BMI than for Blacks, Hispanics, and Whites

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 718 (Actual)
Dates: Start 2007-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in body mass index in adults and body mass index percentile in children. | Baseline to 18 months.
  Height and weight measures will be taken in adults and children to calculate body mass index in adults and body mass index percentile in children.

SECONDARY OUTCOMES:
Change in adiposity for adults and children as measured by change in waist circumference, triceps, and subscapular skinfold measures. | Baseline to 18 months.
  Waist circumference and triceps and subscapular skinfold measures.
Change in health behaviors as measured by nutrition and exercise in adults and children. | Baseline to 18 months.
  nutrition and exercise behaviors in adults and children based on questionnaire scores.
Change in self-efficacy in adults and children as measured by belief that they can improve their eating and exercise behaviors. | Baseline to 18 months.
  eating and exercise self-efficacy in adults and children based on questionnaire scores.

CONTACTS AND LOCATIONS:
Overall Officials: Diane C Berry, PhD, ANP-BC, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Berry DC, McMurray RG, Schwartz TA, Adatorwovor R. Benefits for African American and white low-income 7-10-year-old children and their parents taught together in a community-based weight management program in the rural southeastern United States. BMC Public Health. 2018 Sep 10;18(1):1107. doi: 10.1186/s12889-018-6006-4. PMID 30200925
- [Derived] Berry DC, McMurray RG, Schwartz TA, Hall EG, Neal MN, Adatorwovor R, Adatorwover R. A cluster randomized controlled trial for child and parent weight management: children and parents randomized to the intervention group have correlated changes in adiposity. BMC Obes. 2017 Dec 4;4:39. doi: 10.1186/s40608-017-0175-z. eCollection 2017. PMID 29225899
- [Derived] McMurray RG, Berry DC, Schwartz TA, Hall EG, Neal MN, Li S, Lam D. Relationships of physical activity and sedentary time in obese parent-child dyads: a cross-sectional study. BMC Public Health. 2016 Feb 6;16:124. doi: 10.1186/s12889-016-2795-5. PMID 26851940
- [Derived] Berry DC, McMurray R, Schwartz TA, Skelly A, Sanchez M, Neal M, Hall G. Rationale, design, methodology and sample characteristics for the family partners for health study: a cluster randomized controlled study. BMC Public Health. 2012 Mar 30;12:250. doi: 10.1186/1471-2458-12-250. PMID 22463125